CLINICAL TRIAL: NCT05768425
Title: DIagnostic Biomarkers and Symptoms in Patients With Alzheimer's Disease and Lewy bodY Dementia - DISPLAY
Brief Title: DIagnostic Biomarkers and Symptoms in Patients With Alzheimer's Disease and Lewy bodY Dementia
Acronym: DISPLAY
Status: Active, not recruiting | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Collaborators: Danish Reference Center for Prion Diseases, Rigshospitalet (Unknown); Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Rigshospitalet (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-22046053
Record Dates: First submitted 2023-02-13; First posted 2023-03-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Dementia With Lewy Bodies; Alzheimer Disease; Mild Cognitive Impairment
Keywords: RT-QuIC; Dementia with Lewy bodies; CSF; Saliva; Olfactory mucosa; Urine; Feces; Blood; Skin
MeSH Terms: conditions — Lewy Body Disease; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid, olfactory mucosa, saliva, skin, urine, feces and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dementia with Lewy Bodies (DLB): Mild cognitive impairment (MCI) to moderate dementia with probable DLB No other severe neurological or psychiatric diseases. No alcohol or drug abuse.
  Interventions: Diagnostic Test: Real-time quaking-induced conversion (RT-QuIC); Diagnostic Test: Cognitive test; Diagnostic Test: Motor examination
- Alzheimers disease (AD): MCI to moderate dementia with probable AD. No other severe neurological or psychiatric diseases. No alcohol or drug abuse.
  Interventions: Diagnostic Test: Real-time quaking-induced conversion (RT-QuIC); Diagnostic Test: Cognitive test; Diagnostic Test: Motor examination
- Healthy Controls (HC): Young healthy controls under the age of 40.
  Interventions: Diagnostic Test: Real-time quaking-induced conversion (RT-QuIC); Diagnostic Test: Cognitive test

INTERVENTIONS:
Diagnostic Test: Real-time quaking-induced conversion (RT-QuIC) — RT-QuIC measures the ability of alpha-synuclein (aSyn) to misfold other aSyn proteins and is an amplification technique.
Diagnostic Test: Cognitive test — Minimal Mental State examination (MMSE), Montreal Cognitive Assessment (MoCA)
Diagnostic Test: Motor examination — Unified Parkinsons Rating Scale (UPDRS)
  Groups: Alzheimers disease (AD); Dementia with Lewy Bodies (DLB)

SUMMARY:
This a study to improve diagnosis of dementia with Lewy bodies with RT-QuIC in different biospecimens.

DETAILED DESCRIPTION:
Background. The number of persons living with dementia is increasing in Denmark and worldwide because the population is generally growing older. Dementia with Lewy bodies (DLB) is the second most prevalent etiology among the neurodegenerative diseases that give rise to dementia.

DLB is characterized by many prodromal symptoms years before dementia is evident. Currently, little is known about the course of symptoms in the prodromal phase, and furthermore, the diagnosis of DLB can be clinically challenging, especially in the early stages. A novel technique for the measurement of misfolded alpha-synuclein (aSyn) is Real-Time Quaking-Induced Conversion (RT-QuIC), which may be able to support the diagnostic process.

Objective: Determining which biospecimen alone or in conjunction with other biospecimens can most accurately discriminate patients with DLB from Alzheimer's disease (AD) assessed by RT-QuIC for aSyn.

Design: Cross-sectional case-control study of the diagnostic accuracy of pathological alpha-synuclein assessed by RT-QuIC in different biospecimens (CSF, skin, olfactory mucosa, saliva, feces, and urine) from patients with DLB versus AD.

Patients will also be scored with tests for cognitive function, dysautonomia, and movement disorders.

ELIGIBILITY:
Inclusion criteria for healthy controls (HC):

* Age 18 - 40 years of age
* Able to cooperate as evaluated by the primary investigator (PI)
* Able to give informed consent

Exclusion criteria

* Signs of neurological/psychiatric conditions
* Known genetic neurodegenerative disease in close family

Inclusion criteria for patients with Dementia with Lewy Bodies (DLB):

* Probable DLB (McKeith et al., 2017) or MCI-LB (McKeith et al., 2020)
* Age > 50 years of age
* Able to give informed consent
* Able to cooperate as evaluated by the PI
* MCI, mild or moderate dementia, and MMSE > 18

Exclusion criteria for patients with DLB:

* Patients not able to give informed consent.
* Current alcohol or drug abuse
* Terminal illness
* Diagnosed with major neurological/psychiatric conditions other than DLB.

Inclusion criteria for controls (patients with Alzheimer's disease (AD)):

* Probable AD (McKhann et al., 2011) or MCI-AD (Albert et al., 2011)
* Age > 50 years of age
* Able to give informed consent
* Able to cooperate as evaluated by the PI
* MCI, mild or moderate dementia, and MMSE > 18

Exclusion criteria for controls (patients with AD):

* Patients not able to give consent.
* Current alcohol or drug abuse
* Terminal illness
* Diagnosed with major neurological/psychiatric conditions other than AD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-five patients with probable DLB or mild cognitive impairment with Lewy bodies (MCI-LB) and 25 patients with AD or MCI-AD controls will be included from the memory clinic.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Real-time quaking-induced conversion | 24 months
  Specificity
Diagnostic accuracy of Real-time quaking-induced conversion | 24 months
  Sensitivity
Diagnostic accuracy of Real-time quaking-induced conversion | 24 months
  Area under the curb

SECONDARY OUTCOMES:
Sense of smell | 24 months
  Test with Sniffin Sticks 16, Score 0- 16 points
Dysautonomia | 24 months
  Unified Parkinsons Rating Scale part I 0-52
Motor functions | 24 months
  Unified Parkinsons Rating Scale part III Score range: 0-132
Cognitive function | 24 months
  Montreal Cognitive Assesment (MoCA) Score range: 0-30
Cognitive function | 24 months
  Minimal Mental State Examination (MMSE) Score range: 0-30

CONTACTS AND LOCATIONS:
Overall Officials: Oskar McWilliam, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Kristian S Frederiksen, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Anja H Simmonsen, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Steen G Hasselbalch, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Gunhild Waldemar, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region; Marie Brunn, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Capital Region
Locations (1):
- Danish Dementia Research Centre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No